CLINICAL TRIAL: NCT06536088
Title: The Relationship Between Spatiotemporal Gait Parameters and Imaging-based Characteristics of Femoroacetabular Impingement (FAI) in Symptomatic Individuals
Brief Title: The Relationship Between Gait and Severity of Femoroacetabular Impingement
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: Iayas10
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with Femoroacetabular Impingement: Symptomatic femoroacetabular impingement patients scheduled for hip arthroscopy
  Interventions: Other: Walking assesment
- Control group: Healthy indivicuals without Femoroacetabular Impingement
  Interventions: Other: Walking assesment

INTERVENTIONS:
Other: Walking assesment — Spatiotemporal walking assessments are performed using the Gait Analyzer app (version 0.9.95.0) on a smartphone. Participants who can walk independently without assistance walk a 25-meter path at their normal speed, with the smartphone securely attached to their body above the third lumbar vertebra using a belt. The app records gait velocity, cadence, step time, step length, and vertical center of mass for all participants.

SUMMARY:
In this study, the spatiotemporal gait parameters of symptomatic femoroacetabular impingement (FAI) patients scheduled for hip arthroscopy are evaluated. Radiological measurements, including the Alpha angle (AA), Lateral Center-Edge Angle (LCEA), and Kellgren-Lawrence (KL) osteoarthritis classification, are recorded from patient files. The relationship between these radiological measurements and walking parameters is assessed. Additionally, the spatiotemporal gait parameters of FAI patients are compared with those of a healthy control group.

Walking assessments provide valuable insights into how Femoroacetabular Impingement (FAI) affects movement and aid in evaluating treatment outcomes. Research indicates that individuals with FAI experience reduced hip motion and slower walking speeds. By analyzing spatiotemporal gait parameters-such as gait velocity, cadence, step length, and vertical center of mass-the impact of FAI on walking can be better understood, leading to the development of targeted treatment strategies. The goal is to explore the correlation between these gait parameters and imaging-based FAI characteristics in affected individuals.

DETAILED DESCRIPTION:
Patients and control groups are compared using the paired samples t-test for parametric data and the Wilcoxon signed ranks test for nonparametric data. The relationship between gait parameters and imaging-based FAI characteristics is examined by calculating the Pearson correlation coefficient (r) for parametric data and the Spearman rank correlation coefficient (rho) for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with femoroacetabular impingement scheduled for hip arthroscopy

Exclusion Criteria:

* Severe hip osteoarthritis
* Hip dysplasia
* Previous ipsilateral and/or contralateral hip surgery,
* Any orthopedic or neurologic pathology that may affect gait patterns

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for hip arthroscopy due to Femoroacetabular impingement syndrome at the Department of Orthopedics and Traumatology, Gazi University Faculty of Medicine, along with a healthy control group matched for age and gender, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Gait velocity | Baseline
  Gait velocity, also known as walking speed, is a crucial parameter in spatiotemporal gait analysis. It refers to the rate at which an individual walks over a given distance and is typically measured in meters per second (m/s).
Cadence | Baseline
  Cadence refers to the number of steps a person takes per minute while walking.
Step length | Baseline
  Step length refers to the distance covered between two consecutive footfalls of opposite feet.
Vertical center of mass | Baseline
  The vertical center of mass refers to the vertical position of the body's center of mass during walking. It is the point where the body's mass is considered to be concentrated and it fluctuates as the person moves.

CONTACTS AND LOCATIONS:
Overall Officials: Ulunay Kanatlı, Professor, Study Director — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)